CLINICAL TRIAL: NCT04690530
Title: Cerebal Hemodynamics and Oxygenation in Critically Ill Patients : Characterization and Effects of Therapeutics
Brief Title: Cerebral Hemodynamics and Oxygenation in Critically Ill Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Other Study IDs: 20reamed02
Record Dates: First submitted 2020-12-18; First posted 2020-12-30 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic | interventions — Respiration, Artificial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- patients admitted in medical intensive care unit who require mechanical ventilation and sedation: The main goals of the study are to characterize cerebral hemodynamics and oxygenation as well as to study the effects of therapeutics on it in critically-ill patients. For this purpose, we plan to include all consecutive patients admitted in our medical intensive care unit who require mechanical ventilation and sedation and in whom the attending physician decides to perform one of the studied therapeutics (fluids, vasopressors or inotropes administration, blood transfusion, prone positioning, passive leg raising test, end-expiratory occlusion test) within the first 72h of ventilation onset. Cerebral hemodynamics (cerebral blood flow and cerebral autoregulation) as well as cerebral oxygenation will be non-invasively studied before and after therapeutics.
  Interventions: Procedure: mechanical ventilation; Drug: Sedation

INTERVENTIONS:
Procedure: mechanical ventilation — mechanical vantilation will be performed
Drug: Sedation — sedation wil be performed

SUMMARY:
Critically-ill patients frequently experience marked changes in mean arterial pressure and carbon dioxide partial arterial pressure, the two major determinants of the cerebral blood flow. In addition, many therapeutics (fluids, vasopressors or inotropes administration, blood transfusion, prone positioning...) can influence these two determinants of cerebral blood flow and thus cerebral blood flow, especially in patients with altered cerebral autoregulation. Nevertheless, cerebral hemodynamics and oxygenation, as well as the effects of the different therapeutics on it have been poorly studied in critically-ill patients. In addition, it has been suggested that impaired cerebral blood flow and impaired cerebral microcirculation may be involved in the pathophysiology of septic encephalopathy in patients with sepsis and/or septic shock. In this study, we aimed to characterize and investigate the effects of different therapeutics on cerebral hemodynamics and oxygenation in critically-ill patients.

ELIGIBILITY:
Inclusion Criteria :

* Patients under mechanical ventilation and sedated within the first 72h of ventilation onset
* Indication to one of the studied therapeutics left at the discretion of the attending physician Exclusion criteria
* Age < 18 years
* Pregnancy
* Inability to obtain a Doppler signal
* Medical history or clinical evidence of neurological disease
* Known severe carotid stenosis (>70%)
* Significant cardiac arrhythmias
* Care-limitation decision.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients admitted in our Medical Intensive Care Unit requiring mechanical ventilation and sedation and in whom the attending physician decides to perform one of the studied therapeutics within the first 72h of ventilation onset. Cerebral hemodynamics (cerebral blood flow and cerebral autoregulation) as well as cerebral oxygenation will be non-invasively studied before and after therapeutics.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Cerebral blood flow | Within the first 72 hours of ventilation onset, before and after therapeutics
  Use of transcranial Doppler

SECONDARY OUTCOMES:
Cerebral autoregulation | Within the first 72 hours of ventilation onset, before and after therapeutics
  Use of transcranial Doppler

OTHER OUTCOMES:
Cerebral oxygenation | Within the first 72 hours of ventilation onset, before and after therapeutics
  Use of non-invasive near-infrared spectroscopy (NIRS)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de NICE, Nice, France

IPD SHARING:
Plan to Share IPD: No
no data sharing plan is planned